CLINICAL TRIAL: NCT02175173
Title: Post-marketing Surveillance of Long-term Administration of Inovelon Tablets in Patients With Lennox-Gastaut Syndrome
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: INO01T
Record Dates: First submitted 2014-06-10; First posted 2014-06-26 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2022-11

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Epileptic encephalopathy, Lennox-Gastaut type
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epileptic encephalopathy, Lennox-Gastaut type | interventions — rufinamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- E2080: Children ages >= 4 years: Patients weighing 15.0-30.0 kg: oral daily dose of 200 mg in two divided doses after meals for the first 2 days. The dose will be increased by up to 200 mg/day every two days. The maintenance dose should be 1000 mg/day in two divided doses after meals. The dose can be increased or decreased within a range not exceeding 1000 mg/day, and should be increased by up to 200 mg/day at intervals not less than 2 days. Patients weighing >= 30.1 kg: Adults: oral daily dose of 400 mg in two divided doses after meals for the first 2 days, then increased by up to 400 mg/day every two days. The maintenance dose should be 1800 mg/day for patients weighing 30.1-50.0 kg, 2400 mg/day for patients weighing 50.1-70.0 kg, and 3200 mg/day for patients weighing 70.1 kg or over in two divided doses after meals. Dose can be increased or decreased within a range not exceeding the above maintenance dose, and should be increased by up to 400 mg/day at intervals not less than 2 days.
  Interventions: Drug: Rufinamide

INTERVENTIONS:
Drug: Rufinamide — Administration of Inovelon 100mg or 200mg Tablets
  Other Names: Inovelon Tablet

SUMMARY:
This surveillance's objectives are

1. Unknown adverse reactions
2. Incidences of adverse drug reaction
3. Efficacy during long-term administration
4. Factors considered to have effect to safety and effectiveness
5. Incidences of status epileptics, skin disorders and hyper sensitivity reaction, and central nervous system-related adverse events(ataxia , somnolence and/or dizzy, etc.)

ELIGIBILITY:
All patients with Lennox-Gastaut syndrome and administrated Inovelon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Lennox-Gastaut Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 707 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Investigations on adverse events and adverse drug reactions | Up to 2 years

SECONDARY OUTCOMES:
Frequency of attacks | 12 weeks and every 6 months up to 2years
Overall assessments of the improvement in the seriousness of seizures | 12 weeks and every 6 months up to 2years

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo